CLINICAL TRIAL: NCT02489383
Title: Comparison to Short and Medium-term Effects of Continuous and Interval Aerobic Exercise Training in Improving Aerobic Capacity, Psychosocial Factors and Impact on the Level of Physical Activity in Patients With Asthma Moderate and Severe
Brief Title: Comparison Between Continuous Versus Interval Exercise Training in Asthmatic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Sao Paulo (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Asthmatic exercise training
Record Dates: First submitted 2015-05-12; First posted 2015-07-03 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Asthma
Keywords: Asthma; Continuous Exercise Training; interval Exercise Training; Clinical Control; Inflammation
MeSH Terms: conditions — Asthma; Inflammation | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous Exercise Training (Active Comparator): The interventions of active comparator will be education program and exercise training.
  Interventions: Other: Continuous Exercise Training; Behavioral: Education Program
- Interval Exercise Training (Active Comparator): The interventions of active comparator will be education program and exercise training.
  Interventions: Other: Interval Exercise Training; Behavioral: Education Program

INTERVENTIONS:
Other: Continuous Exercise Training — The continuous training (CT) will be held in two weekly sessions lasting total of 40 minutes and 5 minutes for heating and 5 to slowdown, and the duration will be 24 sessions (3 months). The exercise sessions will be will be performed on a stationary bicycle, with the initial intensity of 70% of VO2max. If the subject sustain continuously training intensity for 2 consecutive sessions without symptoms breathing, exercise intensity will be increased by 5% of heart rate. The patient may stop the activity if he has any symptoms or respiratory distress, returning it as soon present improvement. Throughout the training, will be monitored heart rate and the level of perception subjective effort (modified Borg scale).
  Arms: Continuous Exercise Training
Other: Interval Exercise Training — The interval training (IT) will be held in two weekly sessions. The IT is individualized and will be performed on a stationary bicycle. Training sessions will be performed with total duration of 40 minutes consisting of 5 minutes extender, 30 minutes from the main part (IT), finishing with five minutes back to calm. In the main part (of 5 to 30 minutes), the patient will perform the exercise with high intensity in the first two weeks, the exercise will be conducted with an intensity 80% of maximum capacity obtained in cycle ergometer test and will cycle for 30 seconds followed by a 30 second recovery period. In the 3rd and 4th weeks, the intensity will be increased to 100% of the maximum obtained. After this period, the intensity will be increased by 5% charge.
  Arms: Interval Exercise Training
Behavioral: Education Program — The education program will discuss issues related to asthma and physical activity. Presentations and group discussions will be carried out, including information about asthma pathophysiology, medication and peak flow meter skills, self-monitoring techniques, environmental control, benefits and current recommendations of physical activity.

SUMMARY:
The treatment of asthma is based in clinical control. However, previous studies have been shown that patients that participate of the programs of regular or aerobic continuous exercise training (CT) presented improvements in the physical conditioning, and quality life, as well as decreased the levels of anxiety and depression, reduced the oxide nitric exhaled and leukocyte migration at the airways and reduced the airway hyperresponsiveness. The regular exercise also is important part in the rehabilitation of other lung disease as well as chronic obstructive pulmonary disease (COPD). Additionally, others studies have been shown the effects of high intensity interval training (IT) in the pulmonary rehabilitation of COPD patients, that after performed IT presented reduction of dyspnea, and increase the physical capacity. In this sense, the impact of IT in the asthmatic patients at the present moment is poorly studied, and necessity of the more investigation to prove the efficiency of this training model for asthma patients.

.

DETAILED DESCRIPTION:
The present study will compare the impact of IT and CT in patients with moderate or severe asthma, and investigate what is the most efficient and increases the physical capacity, and quality of life and reduces the inflammatory mediators.

Sixty asthmatic adults will be randomly assigned into two groups: CT (Continuous training) or IT (Interval training). CT will have treatment 2x week, 40 min./session, 60-75% of maximum heart rate intensity and IT also 2x week, 40 min./session, 80-140% of the maximum load intensity, both performed in ergometer cycle by 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Asthma moderate and severe
* Asthma will diagnosed (Global Initiative for Asthma - GINA)
* Body Mass Index (BMI) < 35kg/m2
* Medical Treatment for at least 6 months
* Clinically stable (i.e., no exacerbation or medication changes for at least 30 days)

Exclusion Criteria:

* Cardiovascular, musculoskeletal or other different chronic lung diseases
* Active cancer
* Pregnant
* Smokers

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Endurance test | After 3 months of intervention
  Measurements at isotime: at identical work rates before and after training, heart rate, perception exertion and dyspnea.

SECONDARY OUTCOMES:
Nitric oxide exhaled measurement | Before and after 3 months of intervention
  The level of nitric oxide exhaled (FEno) in the patients with asthma will be quantified with use of the equipment Niox Mino (Niox, Solna, Sweden).
Quantification of Inflammatory mediators | Before and after 3 months of intervention
  The levels of inflammatory mediators interleukin (IL)-4, IL-5, IL-6, IL-8, IL-2, IL-12, IL-17, Interferon gamma (IFN-γ), Tumor necrosis factor alpha (TNF-α), IL-10, and chemokines IL-8, Regulated on Activation, Normal T cell Expressed and Secreted (RANTES), Monocyte Chemoattractant Protein-1 (MCP-1), Monokine induced by gamma interferon (MIG), Interferon gamma-induced protein-10 (IP-10) e Transforming Growing Factor-beta (TGF-b) in the serum will be analyzed by Cytometric bead array (CBA) technique (BD Biosciences, San Jose, California, EUA).
Analysis of cortisol in the serum | Before and after 3 months of intervention
  The level plasmatic of cortisol hormone will be quantified by fluoroimmunoassay by AutoDelfia (Turku, Finland).
Level of physical activity | Before and after 3 months of intervention, and after 3 months of follow up
  The level of Physical activity will be analyzed using a pedometer Yamax model PW 610 (Yamasa, Japan) during 7 consecutive days.
Clinical Control | Before and after 3 months os intervention, ans after 3 months of follow up
  Clinical control will be evaluated by asthma control questionnaire (ACQ)
Health related quality of life | Before and after 3 months os intervention, and after 3 months of follow up
  Health related quality of life will be assessed by Asthma Quality Life Questionnaire (AQLQ)
Level of depression and anxiety | Before and after 3 months os intervention, and after 3 months of follow up
  The symptoms of depression and anxiety will be assessed by Hospital Anxiety and Depression (HAD)
Lung function | Before and after 3 months os intervention, and after 3 months of follow up
  Lung volumes will be assessed by Spirometry
Physical capacity | Before and after 3 months os intervention
  Maximal aerobic capacity (VO2max) will be assessed by Cardiopulmonary exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Celso RF Carvalho, PhD, Principal Investigator — University of São Paulo General Hospital
Locations (2):
- Brazil (2):
  - Physical Therapy, and Clinical Hospital of Sao Paulo University Medical School (HCFMUSP), São Paulo, São Paulo
  - Hospital das Clínicas da Faculadade de Medicina da USP, São Paulo, São Paulo